CLINICAL TRIAL: NCT04997447
Title: Enforced Reduction in Physical Activity and Recovery in Older Adults
Acronym: ENDURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jyvaskyla (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SKR:271901-36456
Record Dates: First submitted 2021-07-01; First posted 2021-08-09 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Muscle Degeneration; Body Weight Changes; Walking, Difficulty
MeSH Terms: conditions — Body Weight Changes; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial, with 2 parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Two weeks of daily step reduction (limited to 2000 steps per day) followed by four weeks of supervised gym-based exercise rehabilitation (twice per week strength training and twice per week cycle endurance training)
  Interventions: Behavioral: Step-reduction/Exercise Rehab
- Control group (No Intervention): Continued monitoring of habitual daily step count without structured intervention. Classic control.

INTERVENTIONS:
Behavioral: Step-reduction/Exercise Rehab — 2-week limited daily steps (<2000), and then 4 weeks of typical strength+endurance exercise for older adults
  Arms: Intervention group

SUMMARY:
Apparently healthy and well-functioning community dwelling 70-80 year-olds will be recruited to the study. All subjects undergo pre-screening for suitability and a physicians examination, as well as 7-day habitual daily steps are measured to ascertain baseline physical activity. Half of the recruited subjects (n=40) will be randomized into the intervention group and half (n=40) randomized into the control group. The intervention group is then required to reduce their daily steps to <2000 for a 2-week period. Thereafter, the intervention group participates to a 4-week strength+endurance training rehabilitation program and no longer has restricted daily step count. The control group continues their normal habitual physical activity level throughout the 6-week study period.

ELIGIBILITY:
Inclusion Criteria:

1. aged 70-80 years,
2. community-dwelling,
3. able to walk 500 m without assistance or use of walking aid and regularly walking >5000 steps per day,
4. MMSE >24,
5. BMI 20-35 kg·m2 (i.e. not underweight or severely obese),
6. no serious cardiovascular or musculoskeletal disease,
7. no risk factors for deep-vein thrombosis (e.g. blood clotting disorder, obesity, bowel diseases, personal or family history of DVT etc.),
8. non-smoker,
9. provision of informed consent.

Exclusion Criteria:

1. Underlying diseases likely to limit lifespan and/or intervention safety. Contraindication for physical exercise or physical tests identified during physician's examination,
2. unwilling/unable to track daily step counts using accelerometer,
3. excessive and regular use of alcohol (more than 7 units per week for women and 14 for men)
4. difficulty in communication due to severe vision or hearing problems
5. unwilling to provide consent or accept randomization into either study group

Ages: 70 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Lean leg mass | 6 weeks
  DXA-measured total lean mass of the legs

SECONDARY OUTCOMES:
Whole-body fat mass | 6 weeks
  DXA-measured total body fat mass
Maximum isometric leg extension force | 6 weeks
  Maximum strength of legs
Walking economy | 6 weeks
  Oxygen uptake while walking at 3 and 5 km.h-1
Short Physical Performance Battery (SPPB) | 6 weeks
  Walking, balance and chair-rise tests
Blood pressure | 6 weeks
  Systolic and diastolic blood pressure during rest (sitting)
HOMA indices | 6 weeks
  Blood glucose and insulin concentration based calculations related to insulin resistance and beta-cell function
White blood cell respiration | 6 weeks
  Isolated white blood cell respiration as a marker for mitochondrial function

CONTACTS AND LOCATIONS:
Overall Officials: Simon Walker, PhD, Principal Investigator — University of Jyväskylä, Finland
Locations (1):
- University of Jyväskylä, Jyväskylä, Central Finland, Finland

IPD SHARING:
Plan to Share IPD: No